CLINICAL TRIAL: NCT03011216
Title: "Ein Training Kognitiver Kontrolle Emotionaler Inhalte im Arbeitsgedächtnis: Effekte Auf Die Häufigkeit Und Auswirkungen Von Grübeln Bei Depressiven Patienten" (English: Training Cognitive Control Over Emotional Information in Working Memory: Effects on the Frequency of Rumination and Its Impact on Mood in the Daily Lives of Depressed Patients)
Brief Title: Effects of Online Cognitive Control Training on Rumination and Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freie Universität Berlin (Other)
Collaborators: University of Stuttgart (Other); University Ghent (Other)
Responsible Party: Principal Investigator, Ulrike Zetsche, Dr. rer. nat., Freie Universität Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZE 1029/3-1
Record Dates: First submitted 2016-12-19; First posted 2017-01-05 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Depression; Rumination - Thoughts
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive emotional cognitive control training (Experimental): Adaptive emotional n-back task: On each trial of this task, participants are presented with an emotional facial expression. Participants have to indicate whether the emotion presented in the current trial is the same as n trials back. In order to train participants at their individual ability level, the n-level varies by trial block based on participants' performance on the previous block.
  The adaptive emotional n-back task is assumed to train the ability to continuously update emotional material in working memory.
  Interventions: Behavioral: Adaptive emotional cognitive control training
- Placebo training (Active Comparator): Adaptive non-emotional feature match task: On each trial of this task, participants are presented with two panels containing 8-12 shapes each. Participants are asked to compare the two panels and decide whether or not they are identical. The panels contain a minimum of 8 shapes and a maximum of 12 shapes, depending on participants' performance on the previous block.
  The adaptive non-emotional feature match task is assumed to train the speed of responding (involving processes like visual search and concentration). It does not trait working memory updating.
  Interventions: Behavioral: Adaptive non-emotional feature match task

INTERVENTIONS:
Behavioral: Adaptive emotional cognitive control training — Is supposed to train ability to continuously update emotional material in working memory.
  Arms: Adaptive emotional cognitive control training
Behavioral: Adaptive non-emotional feature match task — Does not train updating of working memory content; may train reaction time speed, visual search, or concentration abilities.
  Arms: Placebo training

SUMMARY:
The present study examines whether a computerized cognitive control training as compared to a placebo (fake) training will reduce the frequency of depressive rumination in depressed individuals. Rumination has been identified as a major risk factor for the onset and recurrence of depressive episodes and it has been suggested that it is linked to deficits in cognitive control functions. It is thus expected that training cognitive control will reduce the frequency of rumination as well as ameliorate its detrimental effect on negative mood states.

DETAILED DESCRIPTION:
Rumination has been shown to intensify dysphoric mood and is one of the best researched risk factors for the onset and recurrence of depressive episodes. Accumulating evidence suggests that the tendency to ruminate is linked to impairments in cognitive control functions, especially to problems discarding no longer relevant negative material from working memory (=working memory updating).

The aim of the present study is to examine whether training to update emotional material in working memory will have an effect on the frequency of using rumination as well as on the impact of rumination on mood in the daily lives of clinically depressed participants. Participants will be randomly assigned to 10 sessions of either online cognitive control training or an online placebo condition. The ability to update emotional material in working memory will be assessed pre and post training by two computer tasks (close and far transfer tasks). The effects of the training on daily rumination and the dynamics between daily mood and rumination will be assessed pre- and post-training, as well as at 3-months follow-up using ambulatory assessment (via smartphone app). It is expected that individuals in the training as compared to the placebo group will show a greater reduction in rumination frequency as well as a reduction in the negative impact of rumination on mood.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) criteria for a current major depressive episode
* 18-65 years of age
* German native language (due to verbal task requirements)

Exclusion Criteria:

* life time diagnosis of any bipolar or psychotic disorder, or substance dependence
* substance use disorder within past 12 months
* current obsessive-compulsive disorder (OCD) or borderline personality disorder (BPS)
* reporting severe underweight (BMI<18), any neurological disease, severe head injury (e.g. severe concussion), or any brain damage (e.g. due to stroke)
* concurrent psychotherapy during the duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Change in rumination frequency in daily life | from 7-day assessment at pre-training (baseline) to (a) 7-day assessment at post-training (within a week after the end of the training phase), and (b) 7-day assessment at 3-months follow-up
  Rumination frequency is measured by 2 items in the ambulatory assessment. The ambulatory assessment is employed for 7 days pre-training, 7 days post-training (within a week after the end of the training phase), and 7 days at 3-months follow-up with 8 prompts per day during each assessment period
Change in the impact of daily rumination on daily mood | from 7-day assessment at pre-training (baseline) to (a) 7-day assessment at post-training (within a week after the end of the training phase), and (b) 7-day assessment at 3-months follow-up
  The impact of rumination on mood is assessed as the effect of rumination at time t on depressed and positive mood at time t+1 in a multi level model; Time t refers to consecutive assessment points in the ambulatory assessment. The ambulatory assessment is employed for 7 days pre-training, 7 days post-training (within a week after the end of the training phase), and 7 days at 3-months follow-up with 8 prompts per day during each assessment period. Rumination frequency is assessed by two items; depressed and positive mood are each assessed by the average score of two items.

SECONDARY OUTCOMES:
Change in the ability to update emotional material in working memory | from pre-training to post-training (within a week after the end of the training phase)
  Manipulation Check: Measured by two computer tasks (non-adaptive n-back task; modified Sternberg task) in the lab sessions pre- and post-training (=within a week after the end of the training phase). Dependent variables are the differences in accuracy rates and reaction times between the experimental and the control condition in these tasks.
Change in depressed mood and depressive symptoms | from 7-day assessment at pre-training (baseline) to (a) 7-day assessment at post-training (within a week after the end of the training phase), and (b) 7-day assessment at 3-months follow-up
  Depressed mood is assessed by the average score of 2 items in the ambulatory assessment. Ambulatory assessment is employed for 7 days pre-training, 7 days post-training (within a week after the end of the training phase), and 7 days at 3-months follow-up with 8 prompts per day during each assessment period.
  Depressive symptoms are assessed by the Center for Epidemiological Studies - Depression Scale.
Change in levels of disability | from pre-training to post-training (within a week after the end of the training phase)
  Level of disability is assessed by the sum score of the self-report version of the World Health Organization Disability Schedule 2.0 in the lab sessions pre- and post-training (=within 7 days after the end of the training phase)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Zetsche, Dr., Principal Investigator — Freie Universität Berlin
Locations (1):
- Freie Universität Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-individualized data files will be uploaded on Open Science Framework (https://osf.io/) when publications are being prepared
Supporting Information: Study Protocol, Analytic Code
Time Frame: De-individualized data files and the analytic code for each publication will be uploaded on Open Science Framework (https://osf.io/) when the respective publication is prepared. The osf link will be made public as soon as the publication appears online.The data will be accessible as long as osf exists.
Access Criteria: There are no access criteria for reading the code and data. However, if a researcher wants to use the data for further analyses, the researcher has to notify the authors and ask for permission.